CLINICAL TRIAL: NCT02616224
Title: A Study To Observe Treatment Patterns and Outcomes in Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Resource constraints
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29019
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer, HER2 Positive Breast Cancer, Metastatic Breast Cancer, Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with unresectable LA/mBC
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was administered in this study.

SUMMARY:
This observational disease registry is a prospective, national, non-interventional study designed to enroll participants who have received an initial diagnosis of unresectable, locally advanced (LA) or metastatic breast cancer (mBC), up to 6 months prior to registry enrolment. These participants will be prospectively followed for at least 5 years after study enrolment to evaluate their anti-cancer treatments. Data on participants' previous anti-cancer treatments for breast cancer will be collected retrospectively at study entry.

ELIGIBILITY:
Inclusion Criteria:

- Initially diagnosed with HER2-positive unresectable LA/mBC no more than 6 months prior to enrolment, although they can have received anti-cancer treatment during that time

Exclusion Criteria:

There are no exclusion criteria for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have an initial diagnosis of unresectable LA/mBC made up to 6 months prior to registry enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) For Each Anti-Cancer Treatment Regimen | Up to approximately 8 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 8 years
Objective Response Rate (ORR) For Each Anti-Cancer Treatment Regimen | Up to approximately 8 years
Number and Percentage of Participants Receiving Each Unique Treatment Regimen Overall and as First-Line Therapy Versus Second-Line Therapy Versus Subsequent-Line Therapy | Up to approximately 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche